CLINICAL TRIAL: NCT06895811
Title: The Safety and Efficacy Evaluation of Universal PSMA Chimeric Antigen Receptor T Cells in the Treatment of Refractory Castration Resistant Prostate Cancer
Brief Title: Clinical Study of Safety and Efficacy of Universal PSMA CAR- T in Refractory CRPC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Bioray Laboratories (Industry)
Responsible Party: Principal Investigator, Ren Shancheng, Professor, Chief of Urology, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-BRL-302
Record Dates: First submitted 2024-11-12; First posted 2025-03-26 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Prostate Cancer; Castration-resistant Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
Keywords: Prostate cancer; Universal CAR-T; Metastatic Castration-resistant Prostate Cancer; Chimeric Antigen Receptor T cell
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PSMA-UCAR T (BRL-302) (Experimental)
  Interventions: Biological: PSMA-UCAR T (BRL-302)

INTERVENTIONS:
Biological: PSMA-UCAR T (BRL-302) — Three patients will be firstly enrolled at a dose level (DL) of 5.0 × 10^6cells/kg in the DL1 group, following lymphodepleting chemotherapy which will be given under instruction of protocol and investigators' assessment;
  Based on preliminary safety data, efficacy information, and PK/PD parameters obtained at DL1 cohort, the investigator may enroll another three patients in a decreased dose level group of DL-2: 3 × 10^6 cells/kg or DL-1:1 × 10^6 cells/ kg, after thorough discussions between the investigators.

SUMMARY:
This is a single-arm, single-center, open-label clinical trial designed to evaluate the clinical safety and tolerability of different doses of Prostate-Specific Membrane Antigen (PSMA)-Universal Chimeric Antigen Receptor (UCAR) T-lymphocytes (PSMA-UCAR T) for the treatment of patients with refractory castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
This is a single-arm, single-center, open-label clinical trial, which aims to evaluate safety and clinical efficacy of different doses of PSMA-UCAR T (BRL-302) in treating patients with refractory CRPC.

Three patients will be firstly enrolled at a dose level (DL) of 5.0 × 10^6cells/kg in the DL1 group. Based on preliminary safety data, efficacy information, and PK/PD parameters obtained at DL1 cohort, the investigator may enroll another three patients in a decreased dose level group of DL-2: 3 × 10^6 cells/kg or DL-1:1 × 10^6 cells/ kg, after thorough discussions between the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understood and voluntarily signed informed consent for this study;
2. Male, aged 18-80 years;
3. Expected survival of more than 6 months;
4. Metastatic castration-resistant prostate adenocarcinoma (CRPC) patients:

   Have received CRPC standard treatment (such as novel hormone therapies, chemotherapy and radium-223, etc., one or more of the combination therapy) after the diagnosis of CRPC, and is ineffective or progressive :PSA continued rising for 3 months, or bone scan/whole-body MRI/PET-CT showed local recurrence or new metastatic lesions, demonstrating disease progression;
5. PSMA expression in tumor cells was positive in immunohistochemical staining of prostate/metastatic biopsy tissue before enrollment (within 6 months prior to enrollment);
6. ECOG score < 2 ;
7. Virological examination HAV (hepatitis A virus), HBV (hepatitis B virus), HCV (hepatitis C virus), HIV (human immunodeficiency virus), TP (Treponema pallidum) quantitative detection was negative, (antigen and antibody screening method unknown, confirmed by nucleic acid method);
8. Hematological parameters met the following criteria: a. hemoglobin > 100 g/L; b. platelet count > 100 × 10^9/L; c. neutrophils > 1.5 × 10^9/L.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will be excluded:

1. Have received any previous treatment with CAR-T therapy ;
2. Have received any previous treatment that targets PSMA;
3. Tumor pathology suggests a special type of prostate cancer (e.g., neuroendocrine prostate cancer, etc.)
4. Severe mental disorders;
5. Suffered from previous malignancies, except for the following: a. basal cell carcinoma or squamous cell carcinoma after standardized treatment; b. having a primary malignancy, but completely resected, with a complete remission time of ≥ 5 years.
6. Subjects with severe cardiovascular disease; a.New York Heart Association (NYHA) stage III or IV congestive heart failure; b.Myocardial infarction ≤ 6 months prior to enrollment or coronary artery bypass graft (CABG); c.Clinically significant ventricular arrhythmia, or history of unexplained syncope, nonvasovagal or not due to dehydration; d.History of severe non-ischemic cardiomyopathy; e.Decreased left ventricular ejection fraction (LVEF < 55%) as assessed by echocardiogram or multigated acquisition (MUGA) scan, abnormal interventricular septal thickness and atrioventricular size associated with myocardial amyloidosis;
7. Active infectious disease or any major infectious event requiring high grade antibiotics;
8. Organ function in the following abnormalities: a. serum aspartate aminotransferase or alanine aminotransferase > 2.5*Upper Limit of Normal (ULN); CK > ULN; CK-MB > ULN; TnT > 1.5*ULN; b. total bilirubin > 1.5*ULN; c. partial prothrombin time or activated partial thromboplastin time or international normalized ratio > 1.5*ULN in the absence of anticoagulant therapy;
9. Participation in other clinical studies in the past three months or previous treatment with any gene therapy product;
10. Intolerance or hypersensitivity to cyclophosphamide or fludarabine chemotherapy;
11. Unsuitability to participate in this clinical study in the opinion of the investigator.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE V5.0) | Through 6 months after CAR T cell infusion
  Safety assessment: toxicity profile
Cytokine Release Syndrome (CRS) grading post CAR T cell infusion. | Through 6 months after CAR T cell infusion
  Safety assessment: toxicity profile
Safety assessment: dose-limiting toxicity | 28 days after CAR T cell infusion
  Incidence of dose-limiting toxicity (DLT) within 28 days. Dose-limiting toxicity (DLT) is defined as any relevant adverse event that ≥ grade 3 and did not resolve to a grade ≤ grade 2 within 28 days after the first infusion back.

SECONDARY OUTCOMES:
Efficacy assessment: PSA changes | 6 months after CAR T cell infusion
  Prostate-Specific Antigen (PSA) changes assessed by serum PSA measurement (ng/ml).
Efficacy assessment: radiographic Progression-Free Survival (rPFS) | 6 months after CAR T cell infusion
  rPFS is defined as the time between treatment with study drug and the development of imaging progression or death from any cause, whichever occurs first, with imaging progression encompassing the evaluation of progression of primary lesions, non-regional lymph node invasion, soft tissue metastases, and bone metastatic lesions according to RECIST 1.1 and PCWG3 criteria.
6-months Progression-Free Survival (PFS) | 6 months after CAR T cell infusion
  PFS is defined as the time between treatment with study drug and disease progression or death from any cause, whichever occurs first, including biochemical progression or radiographic progression after evaluation according to RECIST 1.1 and PCWG3 criteria according to the included.
Pharmacokinetics (PK) assessment: expansion of CAR T cells | From Day 1 till at least 3 months after CAR T cell infusion
  With the day of the first infusion of the cellular preparation recorded as D0, the monitoring phase of the pharmacokinetic study started from 1 day before the first infusion (D-1).
  Expansion of CAR T cells will be assessed by concentration profile of CAR-T cells in peripheral blood after PSMA-UCAR T infusion.
Pharmacokinetics (PK) assessment: persistence of CAR T cells | From Day 1 till at least 3 months after CAR T cell infusion
  With the day of the first infusion of the cellular preparation recorded as D0, the monitoring phase of the pharmacokinetic study started from 1 day before the first infusion (D-1).
  Persistence of CAR T cells will be assessed by T-cell survival time (area under the curve AUC0-28 at 28 days and area under the curve AUC0-90 at 90 days);
Pharmacodynamics (PD) assessment eg. (Level of IL-6) | From Day 1 till at least 3 months after CAR T cell infusion
  Pharmacokinetic (PD) endpoints is assessed by changes in serum cytokine levels (eg.IL-6) after PSMA-UCAR T infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Shancheng Ren, MD, PhD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Changzheng hospital, Shanghai, Shanghai Municipality, China